CLINICAL TRIAL: NCT03845179
Title: The Blood Glucose-lowering Effect of Glucose-dependent Insulinotropic Polypeptide
Brief Title: GA 6: The Blood Glucose-lowering Effect of Glucose-dependent Insulinotropic Polypeptide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Signe Stensen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18040916
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, cross-over.
Who Masked: Participant, Investigator
Masking Description: Double blinded study. Both participants and investigators are blinded to interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet for placebo treatment period. Following treatment: 2 separate interventions/study days (placebo infusion and GIP receptor antagonist)
  Interventions: Other: Placebo; Other: GIP receptor antagonist; Other: Placebo tablet
- DPP-4 inhibitor (Active Comparator): DPP-4 inhibitor treatment for active treatment period. Following treatment: 2 separate interventions/study days (placebo infusion and GIP receptor antagonist)
  Interventions: Other: Placebo; Other: GIP receptor antagonist; Drug: DPP-4 inhibitor

INTERVENTIONS:
Other: Placebo — Saline infusion
Other: GIP receptor antagonist — Used for infusion on study days
Drug: DPP-4 inhibitor — Oral administration of DPP-4 inhibitor in active treatment period
  Other Names: Sitagliptin
  Arms: DPP-4 inhibitor
Other: Placebo tablet — Oral administration of placebo tablet in placebo treatment period
  Arms: Placebo

SUMMARY:
This study will investigate if the effect of DPP-4 inhibitors is mediated in part by Glucose-dependent insulinotropic polypeptide.

DETAILED DESCRIPTION:
A randomized, placebo controlled study. Using a GIP receptor antagonist, we will investigate the glucose lowering effect of GIP during treatment with DPP-4 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes, treatment: lifestyle changes or metformin
* HbA1c < 75 mmol/mol

Exclusion Criteria:

* diagnosed liver disease
* eGFR < 60 ml/min/1,73m2
* NYHA III or IV
* anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
C-peptide | 5 hours
  Concentrations of C-peptide during GIP receptor antagonism compared to placebo

SECONDARY OUTCOMES:
Plasma glucose | 5 hours
  Concentrations of plasma glucose during GIP receptor antagonism compared to placebo
Insulin | 5 hours
  Concentrations of insulin during GIP receptor antagonism compared to placebo
Total and intact GIP | 5 hours
  Concentrations of total and intact GIP during GIP receptor antagonism compared to placebo
Total and intact GLP-1 | 5 hours
  Concentrations of total and intact GLP-1 during GIP receptor antagonism compared to placebo
Glucagon | 5 hours
  Concentrations of glucagon during GIP receptor antagonism compared to placebo
CTX | 5 hours
  Concentrations of CTX during GIP receptor antagonism compared to placebo
Lipids | 5 hours
  Concentrations of lipids during GIP receptor antagonism compared to placebo

OTHER OUTCOMES:
Gallbladder volume | 5 hours
  Measures from ultrasound sonography
Systolic and diastolic blood pressure | 5 hours
  Repeated measures
heart rate | 5 hours
  Repeated measures

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stensen S, Gasbjerg LS, Rosenkilde MM, Vilsboll T, Holst JJ, Hartmann B, Christensen MB, Knop FK. Endogenous Glucose-Dependent Insulinotropic Polypeptide Contributes to Sitagliptin-Mediated Improvement in beta-Cell Function in Patients With Type 2 Diabetes. Diabetes. 2022 Oct 1;71(10):2209-2221. doi: 10.2337/db22-0059. PMID 35796651